CLINICAL TRIAL: NCT03094221
Title: Clinical Utility and Validation of the Rhythmia Mapping System for the Treatment of Cardiac Arrhythmias
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Elad Anter, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2014P000240
Record Dates: First submitted 2015-10-14; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Cardiac Arrhythmias; Electroanatomic Mapping; Cardiac Ablation
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arrhythmia Mapping: The study sample includes patients referred for three different types of cardiac arrhythmias, which will be the studied categories: 1) atrial flutter/fibrillation, 2) atrial tachycardia, 3) ventricular tachycardia. Patients will undergo standard of care mapping and ablation procedures.
  Interventions: Device: Rhythmia Mapping System

INTERVENTIONS:
Device: Rhythmia Mapping System — Arrhythmia mapping will be performed using the Rhythmia mapping system, including its mapping catheter, either in the atria or ventricles depending on the clinical arrhythmia being treated. Detailed mapping will be performed to determine tissue voltage and arrhythmia mechanism/location according to standard clinical practice. This part of the study will take approximately 90-120 minutes. The catheter position and contact will be visualized with intra-cardiac echocardiography, which is also routinely used during these procedures, and to monitor for potential clinically related complications. Images will be recorded to establish criteria for mapping.

SUMMARY:
The purpose of this study is to compare two different types of three-dimensional electroanatomic mapping systems used for the treatment of cardiac arrhythmias. The systems will be compared in regards to its ability to successfully map and ablate a clinical arrhythmia, as well as the time invested in this activity.

DETAILED DESCRIPTION:
Despite the advancement in catheter ablation technology over the past decade, the essential step in therapy entails identification and accurate mapping of the arrhythmia mechanism and its anatomical substrate. These are performed with the assistance of mapping systems and catheters able to record high fidelity local electrical activity of the heart (electrogram, EGM) and display it in three-dimensional views. Current mapping systems are limited by slow and incomplete arrhythmia mapping, limiting successful therapies.

The Rhythmia™ Mapping System (Rhythmia), including its novel basket catheter (IntellaMap Orion™ High Resolution Mapping Catheter), is an FDA approved mapping system available for use during clinical, standard of care electrophysiology procedures at BIDMC. Its unique design allows improved mapping resolution of cardiac arrhythmias, particularly those with complex disease substrate, such as atrial and ventricular tachycardias. Specifically, the investigators plan to enroll patients undergoing electrophysiology study and ablation for atrial flutter/fibrillation, atrial tachycardia and ventricular tachycardia. The system was developed to provide high-resolution maps based on the rapid, automated acquisition of a very large number of low noise electrograms. This mapping system was designed to improve the speed and clinical outcomes over other systems that do not have this rapid automated acquisition capability.

The Rhythmia mapping system is FDA approved and will be made available for use in clinical procedures at BIDMC. Rhythmia will be installed in one of the three electrophysiology labs at BIDMC and the use of the system is at the discretion of the electrophysiologist performing the procedure. Thus, using or not using the Rhythmia system to guide arrhythmia mapping and ablation is not a deviation from the standard of care.

The goal of this registry study is to examine the clinical utility of the system to create accurate electroanatomical maps and validate the data acquired by comparing it with historical cohorts of electroanatomical signals and their corresponding maps created with the traditional Carto®3 electroanatomic mapping system (Biosense Webster, Inc).

Patients will only be approached for enrollment when the treating physician has elected to utilize the Rhythmia mapping system during the standard clinical procedure. The data acquired will be collected by a member of the research team in a clinical registry for offline analysis.

The aim/hypotheses tested by this study include:

* The Rhythmia mapping system will result in the creation of accurate, high resolution 3D electroanatomical maps, defined as the ability to successfully map the arrhythmia circuit (yes/no) and ablate the arrhythmia (yes/no).
* The time to create an electroanatomical map with the Rhythmia mapping system will be significantly shorter than in historical cohorts using the traditional Carto®3 system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients above the age of 18 years old.
2. Patients with the diagnosis of atrial or ventricular arrhythmias presenting for electrophysiology study.
3. Patients must be able to understand and critically review the informed consent form.

Exclusion Criteria:

1. Patients whom are unable to provide informed consent.
2. Patients with ventricular hypertrophy (LV septum thickness ≥15mm).
3. Patients with prosthetic or stenotic cardiac valves present in the chamber where endocardial mapping is planned
4. Patients with active systemic infections
5. Patients that are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients who present for standard of care catheter ablation procedures for atrial and ventricular arrhythmias.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-01 (Actual)

PRIMARY OUTCOMES:
Arrhythmia Mapping (Yes/No) | Enrollment (Clinical Procedure)
  Ability to successfully map and characterize clinical arrhythmia as confirmed with conventional techniques.
Ablation Success - Elimination of Clinical Arrhythmia (Yes/No) | Enrollment (Clinical Procedure)
  Ability to ablate and eliminate the clinical arrhythmia

SECONDARY OUTCOMES:
Mapping Time (minutes) | Enrollment (Clinical Procedure)
  Mapping time required to characterize the clinical arrhythmia

CONTACTS AND LOCATIONS:
Overall Officials: Elad Anter, MD, Principal Investigator — Beth Israel Deaconess Medical Center, Harvard Medical School
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States